CLINICAL TRIAL: NCT05243238
Title: Hesperidin-Diosmin Effect on Metabolic Syndrome and Diabetic Neuropathy Among Patients With Type 2 Diabetes Mellitus
Brief Title: Hesperidin and Diosmin Effect on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hasnaa Osama, Lecturer of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSU REC FWA#: FWA00015574
Record Dates: First submitted 2022-02-03; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Metabolic Syndrome and Diabetic Neuropathy
MeSH Terms: conditions — Metabolic Syndrome; Diabetic Neuropathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hesperidin group (Active Comparator)
  Interventions: Dietary Supplement: dietary supplement flavonoids
- Diosmin (Active Comparator)
  Interventions: Dietary Supplement: dietary supplement flavonoids
- Hesperidin and diosmin (Active Comparator)
  Interventions: Dietary Supplement: dietary supplement flavonoids
- control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: dietary supplement flavonoids — patients were allocated to receive either hesperidin, diosmin, or combination of both and the fourth group was assigned as a control group without intervention
  Arms: Diosmin; Hesperidin and diosmin; Hesperidin group

SUMMARY:
The components of metabolic syndrome (MetS), particularly obesity and dyslipidemia, are linked to peripheral neuropathy (PN) among patients with diabetes or even without diabetes. Several studies revealed that complementary and herbal medicine could provide a potential for PN management and MetS components. Thus, designing clinical trials with interventions combinations to achieve a considerable improvement is highly recommended. Hesperidin and diosmin, citrus-derived flavonoids, have been reported to possess anti-hyperlipidemic, anti-inflammatory, analgesic, antioxidant, antidiabetic, and anti-hypertensive effect with high tolerability and safety profile

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes adult patients who meet metabolic syndrome criteria and with diabetic neuropathy

Exclusion Criteria:

patients without any parameter of inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
metabolic syndrome components | 12 weeks
  Waist circumference, (cm)
metabolic syndrome components | 12 weeks
  FBG, mg/dl
metabolic syndrome components | 12 weeks
  LDL, mg/dl
metabolic syndrome components | 12 weeks
  HDL
metabolic syndrome components | 12 weeks
  TGs, mg/dl
MNSI score for neuropathy | 12 weeks
  neuropathy improvement if MNSI score decreased

CONTACTS AND LOCATIONS:
Locations (1):
- University, Al Fayyum, Egypt

REFERENCES:
- [Derived] Osama H, Hamed EO, Mahmoud MA, Abdelrahim MEA. The Effect of Hesperidin and Diosmin Individually or in Combination on Metabolic Profile and Neuropathy among Diabetic Patients with Metabolic Syndrome: A Randomized Controlled Trial. J Diet Suppl. 2023;20(5):749-762. doi: 10.1080/19390211.2022.2107138. Epub 2022 Aug 10. PMID 35946912